CLINICAL TRIAL: NCT02732652
Title: Specificity and Sensitivity of Glycosaminoglycan Scores in the Early Diagnosis of Recurrent Renal Cell Carcinoma
Brief Title: Glycosaminoglycan Scores as Monitoring Biomarkers in Confined Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Chalmers University of Technology (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Jens Nielsen, Professor, Chalmers University of Technology
Other Study IDs: GAG-RCC-01
Record Dates: First submitted 2016-03-16; First posted 2016-04-11 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ethylenediaminetetraacetic acid (EDTA)-plasma from blood obtained through venipuncture; and any-void urine
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, a score based on glycosaminoglycan (GAG) profiling in subjects with suspicion of renal cell carcinoma (RCC) is hypothesized to distinguish malignant masses when early actionable clinical decisions are desirable. For example to diagnose early recurrence after surgical treatment; to screen population at risk of RCC; or to distinguish benign masses from RCC before surgical treatment. To this end, plasma and urine GAGs will be measured in a prospective cohort of patients referred to surgical treatment for RCC. The resulting GAG scores are then correlated to post-surgical recurrence, to post-surgical definitive diagnosis and and to tumor size if RCC. In a subset cohort of patients at high risk of RCC recurrence, plasma and urine GAGs will be monitored to observe its correlation with disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for partial or radical nephrectomy for suspicion of renal cell carcinoma
* Predicted life expectancy over 2 months
* Standard imaging evaluation 12 weeks prior to inclusion
* Planned for standard imaging within 16 weeks after start of therapy

Exclusion Criteria:

* Lack of proper compliance to accept continuous samplings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred for partial or radical nephrectomy for suspicion of renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-06; Primary Completion 2021-05 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve (AUC) for the sensitivity/specificity of plasma/urine glycosaminoglycan scores in the prediction of renal cell carcinoma recurrence after surgery | Every 6 or 12 months after surgery up to 5 years
  Radiological assessment of patients with definitive diagnosis of RCC and classified as high risk will be carried out as standard-of-care during follow-up and subjected to correlative analysis relative to the plasma/urine glycosaminoglycan scores (or their change) as assessed by longitudinal sampling.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | Before surgery
  Survival analysis will be performed by Kaplan Meier and significance analysis will use the log-rank test. Cox multivariate analysis will be performed to look at the number and molecular characteristics of the glycosaminoglycan scores as independent prognostic parameters of survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Nielsen, PhD, Principal Investigator — Chalmers University of Technology; Sven Lundstam, M.D. PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be accessible upon study publication

REFERENCES:
- [Result] Gatto F, Dabestani S, Bratulic S, Limeta A, Maccari F, Galeotti F, Volpi N, Stierner U, Nielsen J, Lundstam S. Plasma and Urine Free Glycosaminoglycans as Monitoring Biomarkers in Nonmetastatic Renal Cell Carcinoma-A Prospective Cohort Study. Eur Urol Open Sci. 2022 Jun 29;42:30-39. doi: 10.1016/j.euros.2022.06.003. eCollection 2022 Aug. PMID 35911082
- See also: Related Info — https://doi.org/10.1016/j.euros.2022.06.003